CLINICAL TRIAL: NCT02611167
Title: Pilot Phase I Study of Allogeneic Bone Marrow-Derived Mesenchymal Stem Cell Therapy for Idiopathic Parkinson's Disease
Brief Title: Allogeneic Bone Marrow-Derived Mesenchymal Stem Cell Therapy for Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mya Schiess, Professor and Adriana Blood Chair in Neurology, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-0026
Record Dates: First submitted 2015-11-11; First posted 2015-11-20 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Parkinson's Disease
Keywords: mesenchymal stem cells
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Bone marrow-derived MSC transplantation (1 x 10 6 MSC/kg) (Experimental): Allogeneic bone marrow-derived MSCs will be delivered intravenously.
  Interventions: Biological: Allogeneic bone marrow-derived MSCs (1 x 10 6 MSC/kg)
- Bone marrow-derived MSC transplantation (3 x 10 6 MSC/kg) (Experimental): Allogeneic bone marrow-derived MSCs will be delivered intravenously.
  Interventions: Biological: Allogeneic bone marrow-derived MSCs (3 x 10 6 MSC/kg)
- Bone marrow-derived MSC transplantation (6 x 10 6 MSC/kg) (Experimental): Allogeneic bone marrow-derived MSCs will be delivered intravenously.
  Interventions: Biological: Allogeneic bone marrow-derived MSCs (6 x 10 6 MSC/kg)
- Bone marrow-derived MSC transplantation (10 x 10 6 MSC/kg) (Experimental): Allogeneic bone marrow-derived MSCs will be delivered intravenously.
  Interventions: Biological: Allogeneic bone marrow-derived MSCs (10 x 10 6 MSC/kg)

INTERVENTIONS:
Biological: Allogeneic bone marrow-derived MSCs (1 x 10 6 MSC/kg) — Bone marrow-derived allogeneic MSCs will be delivered intravenously in escalating doses of 1 x 10 6 MSC/kg, 3 x 10 6 MSC/kg, 6 x 10 6 MSC/kg, or 10 x 10 6 MSC/kg of body weight to a population of patients with idiopathic Parkinson's disease (iPD).
  Arms: Bone marrow-derived MSC transplantation (1 x 10 6 MSC/kg)
Biological: Allogeneic bone marrow-derived MSCs (3 x 10 6 MSC/kg) — Bone marrow-derived allogeneic MSCs will be delivered intravenously in escalating doses of 1 x 10 6 MSC/kg, 3 x 10 6 MSC/kg, 6 x 10 6 MSC/kg, or 10 x 10 6 MSC/kg of body weight to a population of patients with idiopathic Parkinson's disease (iPD).
  Arms: Bone marrow-derived MSC transplantation (3 x 10 6 MSC/kg)
Biological: Allogeneic bone marrow-derived MSCs (6 x 10 6 MSC/kg) — Bone marrow-derived allogeneic MSCs will be delivered intravenously in escalating doses of 1 x 10 6 MSC/kg, 3 x 10 6 MSC/kg, 6 x 10 6 MSC/kg, or 10 x 10 6 MSC/kg of body weight to a population of patients with idiopathic Parkinson's disease (iPD).
  Arms: Bone marrow-derived MSC transplantation (6 x 10 6 MSC/kg)
Biological: Allogeneic bone marrow-derived MSCs (10 x 10 6 MSC/kg) — Bone marrow-derived allogeneic MSCs will be delivered intravenously in escalating doses of 1 x 10 6 MSC/kg, 3 x 10 6 MSC/kg, 6 x 10 6 MSC/kg, or 10 x 10 6 MSC/kg of body weight to a population of patients with idiopathic Parkinson's disease (iPD).
  Arms: Bone marrow-derived MSC transplantation (10 x 10 6 MSC/kg)

SUMMARY:
The purpose of this study is to assess the safety, feasibility, and efficacy of intravenous allogeneic bone marrow-derived mesenchymal stem cell (MSC) therapy for idiopathic Parkinson's disease (iPD).

DETAILED DESCRIPTION:
Allogeneic bone marrow-derived mesenchymal stem cells (MSCs) will be delivered intravenously at one of four doses: 1 x 10 6 MSC/kg, 3 x 10 6 MSC/kg, 6 x 10 6 MSC/kg, or 10 x 10 6 MSC/kg of body weight to a population of patients with idiopathic Parkinson's disease (iPD). The infusion will be at 1 week after the baseline visit, following two screening visits. Patients will be followed until 52 weeks after the infusion visit. The safety of the therapy, as well as the impact of the therapy on the rate of Parkinson's disease (PD) progression, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 45 and 70. The 45-year-old age cutoff ensures that we do not enroll juvenile PD patients.
* Diagnosis of Parkinson disease by the United Kingdom (UK) brain bank criteria including the presence of 2 cardinal signs of PD plus bradykinesia. Diagnosis will be confirmed by the PI or other specialists in Movement Disorders and based on medical history, physical and neurological exams. Patients should have an asymmetric onset, unilateral symptoms and a negative pull test. (See Appendix A)
* Moderate to severe microsmia (UPSIT <29).
* A modified Hoehn and Yahr stage of 3 or less in the levodopa OFF state. (See Appendix B)
* Diagnosis of PD between 4 to 7 years.
* Robust response to dopaminergic therapy (defined as greater than 33% reduction in symptoms (on the Unified Parkinson's Disease Rating Scale; UPDRS) when measured in the ON medicine state compared to OFF state.
* If subject is taking any central nervous system acting medications (e.g., benzodiazepines, antidepressants, hypnotics) regimen must be optimized and stable for 90 days prior to the screening visit.
* A stable Parkinson's disease symptomatic therapy for at least 90 days prior to screening and not projected to require additional Parkinson's disease symptomatic therapy for at least one year from the baseline visit.
* Women of childbearing potential will be required to use a reliable form of contraception from 30 days prior to baseline visit until 6 months after the final dose of the study drug.

Exclusion Criteria:

* Atypical or drug-induced Parkinsonism.
* A UPDRS rest tremor score of 3 or greater for any limb.
* A Montreal Cognitive Assessment (MoCA) score of less than 25. (See Appendix C)
* Clinical features of psychosis or refractory hallucinations.
* Uncontrolled seizure disorder, defined as a seizure within the last 6 months.
* Developmental delay.
* Chronic kidney disease defined as glomerular filtration rate (GFR) < 50 mL/min/m2.
* Hepatic disease or altered liver function as defined by alanine transaminase (ALT) >150 U/L and or T. Bilirubin >1.6 mg/dl at admission.
* Presence of clinically refractory orthostatic hypotension at the screening or baseline visit defined as greater than or equal to 20 mmHg change in systolic BP and greater than or equal to 10 mmHg change in diastolic BP from sitting position to standing after 2 minutes that does not respond to medical treatment or baseline sitting BP less than 90/60.
* History of congestive heart failure, clinically significant bradycardia, presence of 2nd or 3rd degree atrioventricular block.
* Pulmonary disease: chronic obstructive pulmonary disease (COPD) with oxygen-requirement at rest or with ambulation; or moderate to severe asthma.
* Active malignancy or diagnosis of malignancy within 5 years prior to the start of screening (Cancer free for at least 5 years is permitted; skin cancers, except for melanoma, are permitted).
* Any diagnosis of autoimmune disease or immunocompromised state, including chemotherapy administration within last 3 years or current immunosuppression as defined by white blood cell (WBC) <3 x 103 cells/ml.
* History of strokes or traumatic brain injury.
* Major surgery within the previous 3 months or planned in the ensuing 6 months.
* Clinically significant abnormalities in the Screening Visit laboratory studies.
* History of use of an investigational drug within 30 days prior to the screening visit.
* History of brain surgery for PD.
* Unable to return for follow-up visits for clinical evaluation, laboratory studies, or imaging evaluation.
* Substance abuse disorder.
* Active anticoagulation treatment.
* Any other condition that the investigator feels would pose a significant hazard to the patient if enrolled or complicate the study assessments.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Safety of allogeneic MSC therapy in patients with iPD as indicated by the presence of adverse events that are confirmed to be related to the therapy | 3 weeks after the first infusion
  Adverse events include renal failure, liver failure, and hemolytic anemia.
Safety of allogeneic MSC therapy in patients with iPD as indicated by the presence of adverse events that are confirmed to be related to the therapy | 12 weeks after the first infusion
  Adverse events include renal failure, liver failure, and hemolytic anemia.
Safety of allogeneic MSC therapy in patients with iPD as indicated by the presence of adverse events that are confirmed to be related to the therapy | 24 weeks after the first infusion
  Adverse events include renal failure, liver failure, and hemolytic anemia.
Safety of allogeneic MSC therapy in patients with iPD as indicated by the presence of adverse events that are confirmed to be related to the therapy | 52 weeks after the first infusion
  Adverse events include renal failure, liver failure, and hemolytic anemia.

SECONDARY OUTCOMES:
Change in motor function as assessed by the Unified Parkinson's Disease Rating Scale (UPDRS) Total score | baseline, 3 weeks
  The UPDRS serves as a disability and impairment scale for progression follow-up and is divided into four sections.
  * Part I: evaluation of mentation, behavior, and mood (13 questions).
  * Part II: evaluation of activities of daily living including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food (13 questions).
  * Part III: motor examination (33 scores based on 18 questions with right, left or other body distributions scores)
  * Part IV: motor complications (6 questions)
  All items have 5 response options with uniform anchors of: 0 = normal, 1 = slight (symptoms/signs with sufficiently low frequency or intensity to cause no impact on function), 2 = mild (symptoms/signs of frequency or intensity sufficient to cause a modest impact on function, 3 = moderate (symptoms/signs sufficiently frequent or intense to impact considerably, but not prevent function), 4 = severe (symptoms/signs that prevent function).
Change in motor function as assessed by the Unified Parkinson's Disease Rating Scale (UPDRS) Total score | baseline, 12 weeks
  The UPDRS serves as a disability and impairment scale for progression follow-up and is divided into four sections.
  * Part I: evaluation of mentation, behavior, and mood (13 questions).
  * Part II: evaluation of activities of daily living including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food (13 questions).
  * Part III: motor examination (33 scores based on 18 questions with right, left or other body distributions scores)
  * Part IV: motor complications (6 questions)
  All items have 5 response options with uniform anchors of: 0 = normal, 1 = slight (symptoms/signs with sufficiently low frequency or intensity to cause no impact on function), 2 = mild (symptoms/signs of frequency or intensity sufficient to cause a modest impact on function, 3 = moderate (symptoms/signs sufficiently frequent or intense to impact considerably, but not prevent function), 4 = severe (symptoms/signs that prevent function).
Change in motor function as assessed by the Unified Parkinson's Disease Rating Scale (UPDRS) Total score | baseline, 24 weeks
  The UPDRS serves as a disability and impairment scale for progression follow-up and is divided into four sections.
  * Part I: evaluation of mentation, behavior, and mood (13 questions).
  * Part II: evaluation of activities of daily living including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food (13 questions).
  * Part III: motor examination (33 scores based on 18 questions with right, left or other body distributions scores)
  * Part IV: motor complications (6 questions)
  All items have 5 response options with uniform anchors of: 0 = normal, 1 = slight (symptoms/signs with sufficiently low frequency or intensity to cause no impact on function), 2 = mild (symptoms/signs of frequency or intensity sufficient to cause a modest impact on function, 3 = moderate (symptoms/signs sufficiently frequent or intense to impact considerably, but not prevent function), 4 = severe (symptoms/signs that prevent function).
Change in motor function as assessed by the Unified Parkinson's Disease Rating Scale (UPDRS) Total score | baseline, 52 weeks
  The UPDRS serves as a disability and impairment scale for progression follow-up and is divided into four sections.
  * Part I: evaluation of mentation, behavior, and mood (13 questions).
  * Part II: evaluation of activities of daily living including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food (13 questions).
  * Part III: motor examination (33 scores based on 18 questions with right, left or other body distributions scores)
  * Part IV: motor complications (6 questions)
  All items have 5 response options with uniform anchors of: 0 = normal, 1 = slight (symptoms/signs with sufficiently low frequency or intensity to cause no impact on function), 2 = mild (symptoms/signs of frequency or intensity sufficient to cause a modest impact on function, 3 = moderate (symptoms/signs sufficiently frequent or intense to impact considerably, but not prevent function), 4 = severe (symptoms/signs that prevent function).
Change in motor function as assessed by the UPDRS Motor score | baseline, 3 weeks
  Parts III and IV of the UPDRS will be performed as described above.
Change in motor function as assessed by the UPDRS Motor score | baseline, 12 weeks
  Parts III and IV of the UPDRS will be performed as described above.
Change in motor function as assessed by the UPDRS Motor score | baseline, 24 weeks
  Parts III and IV of the UPDRS will be performed as described above.
Change in motor function as assessed by the UPDRS Motor score | baseline, 52 weeks
  Parts III and IV of the UPDRS will be performed as described above.
Change in motor function as assessed by Timed-Up-and-Go (TUG) | baseline, 3 weeks
  Time in seconds required to stand from a chair, walk 7meters, turn, walk back to the chair and sit down.
Change in motor function as assessed by Timed-Up-and-Go (TUG) | baseline, 12 weeks
  Time in seconds required to stand from a chair, walk 7meters, turn, walk back to the chair and sit down.
Change in motor function as assessed by Timed-Up-and-Go (TUG) | baseline, 24 weeks
  Time in seconds required to stand from a chair, walk 7meters, turn, walk back to the chair and sit down.
Change in motor function as assessed by Timed-Up-and-Go (TUG) | baseline, 52 weeks
  Time in seconds required to stand from a chair, walk 7meters, turn, walk back to the chair and sit down.
Change in disability as measured by the Modified Hoehn and Yahr Scale | baseline, 3 weeks
  The Modified Hoehn and Yahr Scale is a staging instrument that defines broad categories of motor function in Parkinson's disease, starting at Stage 0: no signs of disease to the highest stage 5: wheelchair bound or bedridden unless aided.
Change in disability as measured by the Modified Hoehn and Yahr Scale | baseline, 12 weeks
  The Modified Hoehn and Yahr Scale is a staging instrument that defines broad categories of motor function in Parkinson's disease, starting at Stage 0: no signs of disease to the highest stage 5: wheelchair bound or bedridden unless aided.
Change in disability as measured by the Modified Hoehn and Yahr Scale | baseline, 24 weeks
  The Modified Hoehn and Yahr Scale is a staging instrument that defines broad categories of motor function in Parkinson's disease, starting at Stage 0: no signs of disease to the highest stage 5: wheelchair bound or bedridden unless aided.
Change in disability as measured by the Modified Hoehn and Yahr Scale | baseline, 52 weeks
  The Modified Hoehn and Yahr Scale is a staging instrument that defines broad categories of motor function in Parkinson's disease, starting at Stage 0: no signs of disease to the highest stage 5: wheelchair bound or bedridden unless aided.
functional connectivity between substantia nigra and dorsal striatum as assessed by resting state functional magnetic resonance imaging (fMRI) | baseline
  Diffusion tensor and T2 imaging with the resting state functional connectivity technique will be used.
perfusion as assessed by arterial spin-labeled (ASL) perfusion MRI | baseline
  Resting cerebral blood flow (CBF) will be measured using a pseudo-continuous arterial spin labeling (pCASL) MRI sequence with gradient-echo echo-planar imaging (EPI), which allows for a non-invasive quantification of CBF.
structural connectivity as assessed by diffusion-weighted MRI for diffusion tensor image (DTI) analysis | baseline
  A set of diffusion-weighted image volumes (32-directions, high angular resolution) will be collected using the gradient overplus option with one B0 (non-diffusion weighted) image volume acquired before the acquisition of one repetition of the diffusion-weighted scans. Diffusion tensor and associated computations will be performed. White matter microstructure will be examined, which represents the structural pathways linking specific cortical and subcortical regions. It will be determined whether there is increased fractional anisotropy and decreased mean diffusivity along white matter fibers that link regions exhibiting increased functional connectivity, such as substantia nigra and dorsal striatum.
volume of subcortical structures as assessed by T1- and T2- weighted MRI with Fluid Attenuated Inversion Recovery | baseline
  Anatomical imaging allows visualization of the brain structure at the level of about 1 cubic millimeter. These scans will be used to estimate the volume of subcortical structures (e.g., putamen, caudate nucleus).
cortical thickness as assessed by T1- and T2- weighted MRI with Fluid Attenuated Inversion Recovery | baseline
  Anatomical imaging allows visualization of the brain structure at the level of about 1 cubic millimeter. These scans will be used to measure cortical thickness (e.g., gray matter density).
Change in gross brain structure as assessed by T1- and T2- weighted MRI with Fluid Attenuated Inversion Recovery | baseline
  Anatomical imaging allows visualization of the brain structure at the level of about 1 cubic millimeter. These scans will be used to detect any gross structural changes or inflammation that appear during the course of treatment.
Change in brain activity as assessed by task state fMRI | baseline
  Whole-brain echo-planar imaging (EPI) runs sensitive to BOLD contrast will be acquired while participants do self-paced finger tapping using their left and right hands at separate points in time, and during the resting state after being instructed to remain still and fixate on a white crosshair displayed on a black background during the functional acquisition. Functional imaging will be done in the OFF medication state. It will be determined whether there is a reduction in the abnormally high activity pattern in motor cortex and an increase in putamen activity.
Change in quality of life as assessed by the modified Schwab and England activities of daily living (ADL) score | baseline, 3 weeks
  The Schwab & England scale is a physician assessment of the subject's level of independence. The subject will be scored on a percentage scale reflective of his/her ability to perform acts of daily living in relation to what he/she did before Parkinson disease appeared. Scores range from 100% to 0% in increments of 10%, where 100% is completely independent and 0% is only vegetative functions.
Change in quality of life as assessed by the modified Schwab and England activities of daily living (ADL) score | baseline, 12 weeks
  The Schwab & England scale is a physician assessment of the subject's level of independence. The subject will be scored on a percentage scale reflective of his/her ability to perform acts of daily living in relation to what he/she did before Parkinson disease appeared. Scores range from 100% to 0% in increments of 10%, where 100% is completely independent and 0% is only vegetative functions.
Change in quality of life as assessed by the modified Schwab and England activities of daily living (ADL) score | baseline, 24 weeks
  The Schwab & England scale is a physician assessment of the subject's level of independence. The subject will be scored on a percentage scale reflective of his/her ability to perform acts of daily living in relation to what he/she did before Parkinson disease appeared. Scores range from 100% to 0% in increments of 10%, where 100% is completely independent and 0% is only vegetative functions.
Change in quality of life as assessed by the modified Schwab and England activities of daily living (ADL) score | baseline, 52 weeks
  The Schwab & England scale is a physician assessment of the subject's level of independence. The subject will be scored on a percentage scale reflective of his/her ability to perform acts of daily living in relation to what he/she did before Parkinson disease appeared. Scores range from 100% to 0% in increments of 10%, where 100% is completely independent and 0% is only vegetative functions.
Change in quality of life as assessed by the Parkinson's Disease Questionnaire (PDQ-39) | baseline, 3 weeks
  The PDQ-39 is a 39 questions Parkinson's Disease self-completed questionnaire that comprises 8 domains: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items) and bodily discomfort (3 items). All items are assumed to impact QoL and must be answered to compute scores for each dimension. Questions are answered based on experiences from the preceding month using a 5-point ordinal scoring system: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, 4 = always. Each scores range from 0 = never have difficulty to 100 = always have difficulty.
Change in quality of life as assessed by the Parkinson's Disease Questionnaire (PDQ-39) | baseline, 12 weeks
  The PDQ-39 is a 39 questions Parkinson's Disease self-completed questionnaire that comprises 8 domains: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items) and bodily discomfort (3 items). All items are assumed to impact QoL and must be answered to compute scores for each dimension. Questions are answered based on experiences from the preceding month using a 5-point ordinal scoring system: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, 4 = always. Each scores range from 0 = never have difficulty to 100 = always have difficulty.
Change in quality of life as assessed by the Parkinson's Disease Questionnaire (PDQ-39) | baseline, 24 weeks
  The PDQ-39 is a 39 questions Parkinson's Disease self-completed questionnaire that comprises 8 domains: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items) and bodily discomfort (3 items). All items are assumed to impact QoL and must be answered to compute scores for each dimension. Questions are answered based on experiences from the preceding month using a 5-point ordinal scoring system: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, 4 = always. Each scores range from 0 = never have difficulty to 100 = always have difficulty.
Change in quality of life as assessed by the Parkinson's Disease Questionnaire (PDQ-39) | baseline, 52 weeks
  The PDQ-39 is a 39 questions Parkinson's Disease self-completed questionnaire that comprises 8 domains: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items) and bodily discomfort (3 items). All items are assumed to impact QoL and must be answered to compute scores for each dimension. Questions are answered based on experiences from the preceding month using a 5-point ordinal scoring system: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, 4 = always. Each scores range from 0 = never have difficulty to 100 = always have difficulty.
Change in cognitive function as assessed by the Montreal Cognitive Assessment (MoCA) | baseline, 52 weeks
  The Montreal Cognitive Assessment is a rapid screening instrument for working memory, visual-spatial abilities, executive function, attention, concentration, language and orientation. The total score ranges from 0 to 30; a score of 26 or above is considered normal.
Change in immunologic response as assessed by plasma concentrations of cytokines | baseline, 3 weeks
  Investigators will assess cytokines associated with inflammation [interleukin-6 (IL-6), Interleukin-1 beta (IL-1β), Tumor Necrosis Factor beta (TNFβ)]; cell growth and differentiation [Brain-derived neurotrophic factor (BDNF), Granulocyte-macrophage colony-stimulating factor (GM-CSF)]; monocyte migration [Fractalkine, Eotaxin, monocyte chemotactic protein 1 (MCP-1), Macrophage Inflammatory Protein 1 beta (MIP-1β)]; and adaptive immune response [interleukin 12 subunit beta (IL-12p40), interleukin 7 (IL-7), interleukin 9 (IL-9), interleukin 4 (IL-4)] will be measured.
Change in immunologic response as assessed by plasma concentrations of cytokines | baseline, 12 weeks
  Investigators will assess cytokines associated with inflammation [interleukin-6 (IL-6), Interleukin-1 beta (IL-1β), Tumor Necrosis Factor beta (TNFβ)]; cell growth and differentiation [Brain-derived neurotrophic factor (BDNF), Granulocyte-macrophage colony-stimulating factor (GM-CSF)]; monocyte migration [Fractalkine, Eotaxin, monocyte chemotactic protein 1 (MCP-1), Macrophage Inflammatory Protein 1 beta (MIP-1β)]; and adaptive immune response [interleukin 12 subunit beta (IL-12p40), interleukin 7 (IL-7), interleukin 9 (IL-9), interleukin 4 (IL-4)] will be measured.
Change in immunologic response as assessed by plasma concentrations of cytokines | baseline, 24 weeks
  Investigators will assess cytokines associated with inflammation [interleukin-6 (IL-6), Interleukin-1 beta (IL-1β), Tumor Necrosis Factor beta (TNFβ)]; cell growth and differentiation [Brain-derived neurotrophic factor (BDNF), Granulocyte-macrophage colony-stimulating factor (GM-CSF)]; monocyte migration [Fractalkine, Eotaxin, monocyte chemotactic protein 1 (MCP-1), Macrophage Inflammatory Protein 1 beta (MIP-1β)]; and adaptive immune response [interleukin 12 subunit beta (IL-12p40), interleukin 7 (IL-7), interleukin 9 (IL-9), interleukin 4 (IL-4)] will be measured.
Change in immunologic response as assessed by plasma concentrations of cytokines | baseline, 52 weeks
  Investigators will assess cytokines associated with inflammation [interleukin-6 (IL-6), Interleukin-1 beta (IL-1β), Tumor Necrosis Factor beta (TNFβ)]; cell growth and differentiation [Brain-derived neurotrophic factor (BDNF), Granulocyte-macrophage colony-stimulating factor (GM-CSF)]; monocyte migration [Fractalkine, Eotaxin, monocyte chemotactic protein 1 (MCP-1), Macrophage Inflammatory Protein 1 beta (MIP-1β)]; and adaptive immune response [interleukin 12 subunit beta (IL-12p40), interleukin 7 (IL-7), interleukin 9 (IL-9), interleukin 4 (IL-4)] will be measured.
Change in suicidal ideation or behaviors as assessed by and Columbia Suicide Severity Rating Scale (CSSRS) | Screening, 3 weeks, 12 weeks, 24 weeks, 52 weeks
  The CSSRS rating scale is a set of questions directed towards eliciting verbalization of suicidal feelings or actions

CONTACTS AND LOCATIONS:
Overall Officials: Mya Schiess, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No